CLINICAL TRIAL: NCT06058559
Title: Effect of Sunflower Lecithin Supplementation on Meibomian Gland Function in Adults With Dry Eye Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: George Washington University (Other)
Collaborators: Virginia Lions Institute Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 101
Record Dates: First submitted 2023-09-22; First posted 2023-09-28 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Dry Eye Disease; Meibomian Gland Dysfunction
MeSH Terms: conditions — Dry Eye Syndromes; Meibomian Gland Dysfunction | interventions — Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sunflower Lecithin (Experimental): Total 4800 mg sunflower lecithin per day taken in 4 softgel capsules
  Interventions: Dietary Supplement: Sunflower lecithin
- Olive Oil (Placebo Comparator): Total 4000 mg olive oil per day taken in 4 softgel capsules
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Sunflower lecithin — Lecithins are a group of essential phospholipids that are involved in a number of biological functions such as lipid-cholesterol transport, transmembrane signaling, and neurological function
  Arms: Sunflower Lecithin
Dietary Supplement: Olive oil — Extra virgin olive oil
  Arms: Olive Oil

SUMMARY:
This prospective study will evaluate the effect of oral sunflower lecithin dietary supplementation on meibomian gland function in adults with dry eye disease.

DETAILED DESCRIPTION:
Enrolled patients in the active arm of the study (n=20) will receive a daily dose of four sunflower lecithin 1,200 mg soft-gel capsules for a duration of 90 days. Patients in the control arm (n=10) will receive four doses of a 1,000 mg placebo soft-gel capsules (containing olive oil). Patients will be evaluated for meibomian gland function and signs and symptoms of dry eye at baseline and at the end of the study using a standardized eye dryness survey (SPEED survey), Tear Breakup Time Measurement, Meibomian Gland Score, and a rapid in-office assessment of years (InflammaDry).

ELIGIBILITY:
Inclusion Criteria:

* Age greater than18 at the time of informed consent
* Clinical diagnosis of dry eye in both eyes
* Fluorescein tear film break-up time (TBUT) less than 10s in both eyes
* The presence of lid margin scaling, telangiectasia, collarette or meibomian gland plugging on slit-lamp examination
* Best-corrected visual acuity (BCVA, Snellen) of 20/40 or better in each eye
* Patient Evaluation of Eye Dryness (SPEED) questionnaire score >6 to <14
* Must understand; be willing and able, and likely to fully comply with study procedures, visit schedule, and restrictions

Exclusion Criteria:

* Any pre-existing ocular disease other than dry eye disease
* Patients with inability to swallow soft gel capsules
* Severe illness, pregnancy or breastfeeding, smoking, and regular use of strongly anticholinergic drugs.
* Drastic change of food and/or food supplements within the last month.
* Other food supplement with fatty acids
* Evidence of acute ocular infection and⁄or intraocular inflammation within 1 month prior to the onset of this study.
* Ocular surgery within the last 6 months.
* Patients treated with topical ocular, steroidal or non-steroidal, anti-inflammatory treatment within the last month.
* Occlusion therapy with lacrimal or punctum plugs within the last 3 months.
* Alterations of the lacrimal drainage system
* Eyelid abnormalities
* Patients on oral tetracycline or corticosteroids
* Active allergy or infection at the ocular surface

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2023-06-20 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of the SPEED questionnaire score at Day 90 | 90 days
  To assess the improvement of dry eye symptoms by SPEED questionnaire. 0 score is the minimum (no dry eye symptom); 64 is the maximum score (most symptomatic). Change = (Day 90 score - Baseline score)

SECONDARY OUTCOMES:
Change from Baseline of Fluorescein Tear Break-Up Time (Seconds) at Day 90 | 90 days
  Fluorescein Tear Break-Up Time (TBUT) is a measurement in seconds of tear film stability. The shorter the TBUT, the lower the tear film stability. Lower tear film stability is associated with dry eye. Change = (Day 90 value - Baseline value)
Change in number of MMP-positive eyes at Day 90 | 90 days
  InflammaDry is a noninvasive immunoassay for detecting the presence of MMP-9 in tears.
Least Squares Mean Change from Baseline in Meibomian Gland Score (MGS) at Day 90 | 90 days
  Meibomian glands on the eyelids assessed by the examiner using a Meibomian Gland Evaluator (MGE) and a slit lamp microscope. An MGE instrument applies a standardized force simulating the pressure of a deliberate blink allowing eye care professionals to observe meibomian gland functionality through a slit lamp. 5 glands in 1 zone (nasal) evaluated for each eye and scored from 0 to 3, with a resultant overall score (MGS) of 0 to 15 for each eye. Scoring as follows: 0 = no secretion (worst), 1 = inspissated, 2 = cloudy, 3 = clear liquid (best). A higher change from baseline score indicates an improvement in meibomian gland function.

CONTACTS AND LOCATIONS:
Overall Officials: David Belyea, MD, Study Chair — The George Washington University
Locations (1):
- The GW Medical Faculty Associates, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No